CLINICAL TRIAL: NCT00451490
Title: The Effect of Agomelatine or Fluoxentine on Heart Rate Variability in Patients With Major Depressive Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study not get the approval by the drug company
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 200610027R
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2007-01

CONDITIONS: Depressive Disorder, Major
Keywords: agomelatin; prozac; heart rate variability; major depression; sleep; depressive symptoms
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — agomelatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Agomelatine
Drug: Fluoxentine

SUMMARY:
Phase advance of HRV will be anticipated in agomelatine group. It is anticipated that both agomelatine and floxentine will increase HRV at the end of the treatment.

DETAILED DESCRIPTION:
Phase advance of HRV will be anticipated in agomelatine group. It is anticipated that both agomelatine and floxentine will have equal efficacy in improvement of depressive symptoms and increasement of HRV at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Asian patients
* Male or female
* 18 to 65 years outpatients
* DSM-IV-TR criteria for Major Depressive Disorder

Exclusion Criteria:

* Patients with cardiac conditions and other physical conditions contraindicated for drug study
* Shift worker
* Patients known to be non-responders to fluoxetine treatment
* Pregnancy, or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-10; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
the Pittsburgh Sleep Quality Index
the Leeds Sleep Evaluation Questionnaire

SECONDARY OUTCOMES:
heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chih Tseng, MD, Principal Investigator — National Taiwan Univetsity Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan